CLINICAL TRIAL: NCT05395975
Title: Assessment of Different Preoxygenation Methods With Oxygen Reserve Index In Cesarean Section
Brief Title: Different Preoxygenation Methods In Cesarean Section
Status: Completed | Type: Observational
Sponsor: Zonguldak Bulent Ecevit University (Other)
Responsible Party: Sponsor
Other Study IDs: 2020/22-24
Record Dates: First submitted 2022-05-12; First posted 2022-05-27 (Actual); Last update posted 2022-05-27 (Actual); Status verified 2020-11

CONDITIONS: Hypoxia; Hyperoxia
Keywords: Oxygen Reserve Index; Preoxygenation; General Anesthesia; Cesarean Section
MeSH Terms: conditions — Hypoxia; Hyperoxia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group I: Preoxygenation with 100% oxygen for 3 minutes
  Interventions: Device: Oxygen Reserve Index
- Group II: 4 deep breaths with 100% oxygen in 30 seconds
  Interventions: Device: Oxygen Reserve Index

INTERVENTIONS:
Device: Oxygen Reserve Index — It is a new non-invasive and continuous measurement parameter that aims to provide information about the oxygen status of patients in the moderately hyperoxic range (100 mmHg< PaO2 ≤ 200 mmHg).

SUMMARY:
The study aimed to evaluate different preoxygenation methods (tidal volume for 3 minutes and 4 deep breaths) in pregnant women with oxygen reserve index (ORI).

After the routine monitoring of healthy ASA II pregnant patients between the ages of 18-45, different preoxygenation methods will be applied, and the oxygen status of the patients will be compared with ORI monitoring.

ELIGIBILITY:
Inclusion Criteria:

* The average operation time is 30 minutes-1.5 hours.
* ASA II risk class
* All pregnant women with a gestational week >36

Exclusion Criteria:

* preeclampsia
* eclampsia
* fetal distress
* morbid obesity
* a history of malignant hyperthermia
* opioid sensitivity
* alcohol or drug addiction
* congestive heart failure
* chronic obstructive pulmonary disease
* coronary artery disease
* anemia, liver and kidney disease
* hypovolemia, hypotension, sepsis
* Those who are allergic to the drugs used in the study and who are suspected of difficult intubation

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients aged 18-45 who had cesarean section under general anesthesia
Sampling Method: Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2021-12-27 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Preoxygenation Methods | During the surgery
  Effects of Different Preoxygenation Methods on SaO2, FiO2 and FeO2 with Oxygen Reserve Index

CONTACTS AND LOCATIONS:
Locations (1):
- Zonguldak Bülent Ecevit University Faculty of Medicine, Zonguldak, Kozlu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes